CLINICAL TRIAL: NCT04495972
Title: Novel Intestinal Microbiota-based Product for Preventing Type 2 Diabetes Mellitus
Brief Title: Intestinimonas for Prevention of Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Caelus Pharmaceuticals BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DM Prevent POC
Record Dates: First submitted 2020-07-27; First posted 2020-08-03 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: PreDiabetes
Keywords: Prediabetic State; Metabolic Syndrome
MeSH Terms: conditions — Prediabetic State; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm: Intestinimonas (Active Comparator): Intestinimonas in capsules
  Interventions: Dietary Supplement: Intestinimonas-capsules
- Placebo arm: Placebo (Placebo Comparator): Placebo in capsules
  Interventions: Dietary Supplement: Placebo-capsules

INTERVENTIONS:
Dietary Supplement: Intestinimonas-capsules — Capsules containing microbiota (Intestinimonas)
  Arms: Experimental arm: Intestinimonas
Dietary Supplement: Placebo-capsules — Placebo capsules are identical to the active treatment
  Arms: Placebo arm: Placebo

SUMMARY:
The study aims to assess the effects of a microbiota-based product containing Intestinimonas in adults with pre-diabetes. The purpose is to determine the safety and efficacy of the microbiota-based product on insulin sensitivity in a target group of prediabetic individuals. In particular, the objective is to evaluate whether Intestinimonas is able to improve the insulin sensitivity, the response to the oral glucose tolerance test (OGTT) and whether it is able to modulate the microbiota composition in the study subjects.

DETAILED DESCRIPTION:
The study aims to assess the effects of a microbiota-based product containing Intestinimonas in adults with pre-diabetes.

Intestinimonas is an aerobic microorganism which produces butyrate and interacts with the local microbiota in small and large intestine.

In preclinical studies, it was demonstrated that the insulin sensitivity can be enhanced by Intestinimonas and similar microbiota.

The purpose is to determine the safety and efficacy of the microbiota-based product on insulin sensitivity in a target group of prediabetic individuals.

The study participants will be subjects who are overweight and are at risk of developing Type 2 diabetes.

The key objective of this randomized, placebo-controlled study is to evaluate whether Intestinimonas is able to improve the insulin sensitivity, to assess the response to the oral glucose tolerance test (OGTT) and whether it is able to modulate the microbiota composition in the study subjects.

Furthermore, in a open-label follow-up of 14 weeks the effect of a high-dose of Intestinimonas will be compared with the low-dose tested in the initial double-blind Randomised Controlled Trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* increased BMI > 25,
* Fasting Plasma Glucose (FPG) 100-125 mg/dl or glucose > 140 after OGTT, or HbA1c 5.7% - 6.4%

Exclusion Criteria:

* Type 2 diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 12 weeks
  as measured by Homeostatic Model Assessment (HOMA) - index

SECONDARY OUTCOMES:
Concentration of Fasting glucose | 12 weeks
  as measured by Glucose in plasma
Level of 2-hour blood glucose Area Under the Curve (AUC) | 12 weeks
  as measured by standard Oral Glucose Tolerance Test (OGTT)

CONTACTS AND LOCATIONS:
Locations (1):
- University Piemonte Orientale, Vercelli, Italy